CLINICAL TRIAL: NCT01902771
Title: A Phase I Study of Dendritic Cell Vaccine Therapy With In Situ Maturation for Pediatric Brain Tumors
Brief Title: Dendritic Cell Vaccine Therapy With In Situ Maturation in Pediatric Brain Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: Edward Ziga (Other)
Responsible Party: Sponsor-Investigator, Edward Ziga, Assistant Professor of Clinical Pediatrics, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130136
Record Dates: First submitted 2013-07-16; First posted 2013-07-18 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Glioma; Brain Cancer; Brain Tumor; Glioblastoma Multiforme; High Grade Glioma
Keywords: Dendritic Cell Vaccine; DCV; Pediatric; Brain Tumor; In Situ; Lysate; Tumor Lysate; Glioblastoma Multiforme; GBM; Pheresis; Leukapheresis; High Grade Glioma; HGG
MeSH Terms: conditions — Glioma; Brain Neoplasms; Glioblastoma | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; Imiquimod; Leukapheresis; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DC Vaccine + Lysate (Experimental): * Leukapheresis: Baseline, post-surgery;
  * Dendritic Cell Vaccine (DC Vaccine): Post-Leukapheresis, administered intradermally once weekly via intradermal injection, for 4 weeks for a total of four vaccinations;
  * Tumor Lysate (Lysate): Post-DC Vaccine therapy. Administered intradermally during weeks 8, 12, 16, and 28;
  * Imiquimod: Self-applied topically by subject before and after scheduled DC Vaccine or Lysate administrations.
  Interventions: Biological: Dendritic Cell Vaccine; Biological: Tumor Lysate; Other: Imiquimod; Procedure: Leukapheresis

INTERVENTIONS:
Biological: Dendritic Cell Vaccine — Post-Leukapheresis. Subjects will receive DC Vaccine administered once weekly, via intradermal injection, for 4 weeks for a total of four vaccinations, per study protocol.
  Other Names: DC Vaccine
Biological: Tumor Lysate — Post-DC Vaccine therapy. Up to 1.5 mg of Lysate of tumor per dose administered via intradermal injection at intervals defined by study protocol.
  Other Names: Tumor Cell Lysate; Lysate of Tumor
Other: Imiquimod — Subjects will self-apply Imiquimod topically to each designated vaccine site before and after scheduled administrations of DC Vaccine or Lysate, per study protocol.
  Other Names: Aldara
Procedure: Leukapheresis — Baseline, post-surgery. Subjects will undergo leukapheresis procedure during baseline, after recovery from surgery to collect peripheral blood mononuclear cells (PBMCs) from which dendritic cells will be obtained, per study protocol.
  Other Names: Pheresis

SUMMARY:
DC vaccine manufactured and partially matured using our standard operating procedures, developed in collaboration with the HGG Immuno Group, then administered through imiquimod treated skin will be safe and feasible in children with refractory brain tumors. This will result in anti-tumor immunity that will prolong survival of subjects treated and results will be consistent with the outcomes found for subjects treated by HGG Immuno Group investigators. Study treatment will correlate with laboratory evidence of immune activation. Correlative studies will also reveal targets in the immune system which can be exploited to improve response for patients on successor trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 1 year and ≤ 29 years
2. Relapse or progression of any central nervous system tumor initially diagnosed before the age of 21 years.
3. Total or subtotal resection of tumor mass, confirmed by assessment by the neurosurgeon and by postoperative MRI scan within 72 hours after surgery. The post-operative assessment should demonstrate residual tumor less than or equal to 2 cm^3 as judged by surgeon or on MRI the tumor should only show linear contrast enhancement at the border of the resection cavity or nodule less than 2 cm^3.
4. No radiotherapy and/or chemotherapy received for at least 1 month before first DC vaccination is to be administered.
5. No treatment with corticosteroids or salicylates for at least 1 week before first vaccination.
6. Life expectancy ≥ 3 months
7. Written consent by patient or parent(s) (if patient is < 18 years) on an institutional review board (IRB)-approved informed consent form prior to any study-specific evaluation. Assent is required from children as per University of Miami (UM) IRB guidelines. Subject must be capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent.
8. Adequate organ function (to be measured at enrollment)

   * Absolute neutrophil count (ANC) ≥750/L
   * Lymphocytes ≥ 500/L
   * Platelets ≥ 75,000/L
   * Hemoglobin ≥ 9 g/dL
   * Aspartate aminotransferase (AST)/Alanine transaminase (ALT) ≤ 2.5 X upper limit of normal (ULN); if liver metastases, ≤ 5 X ULN
   * Serum Creatinine ≤ 1.5 X ULN
   * Total Bilirubin ≤ 3 X ULN
   * Albumin > 2 g/dL
9. Subjects must agree to use adequate method of contraception or abstinence throughout and up to 4 weeks after the study treatment completion.
10. Karnofsky score ≥ 70 or Eastern Cooperative Oncology Group (ECOG) status of 0 or 1.

Exclusion Criteria:

1. Pregnancy.
2. Breast feeding females.
3. Any concomitant participation in other therapeutic trials.
4. Virus serology positive for HIV (testing is not required in the absence of clinical suspicion).
5. Documented immunodeficiency or autoimmune disease.
6. Other active malignancies.
7. Refusal to use adequate contraception for fertile patients (females and males) during the study and for 30 days after the last dose of study treatment.
8. Any serious or uncontrolled medical or psychiatric condition that in the opinion of the investigator makes the patient not able to participate in the study.
9. Application of gliadel wafers within the prior 4 months or a plan to place Gliadel wafers at the time of resection for tumor acquisition for study.

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
Rate of Toxicity in Study Participants Receiving Protocol Therapy | Up to 28 Weeks
  Rate of treatment-limiting toxicities (TLT) and/or adverse events in study participants receiving protocol therapy.
Rate of Feasibility of Protocol Therapy in Study Participants | Up to 4 Weeks
  Rate of feasibility of protocol therapy in study participants. Feasibility refers to clinical feasibility - whether or not the patient can have enough monocytes removed to manufacture Dendritic Cells.

SECONDARY OUTCOMES:
Rate of Prolonged Survival or Prolonged Progression-Free Survival in Study Participants | Up to 24 Months
  Rate of prolonged survival or prolonged progression-free survival in study participants. Overall Survival is defined as the time elapsed from the start of treatment until death. For surviving patients, follow-up will be censored at the date of last contact. Progression-Free Survival (PFS) is defined as the time elapsed from the start of treatment to the date of documented progression or death, whichever comes first.
Rate of Measurable Immune Response in Subjects Receiving Protocol Therapy. | Up to 24 months
  Rate of measurable immune response in subjects receiving protocol therapy demonstrated by measurement levels of Myeloid Derived Suppressor Cells before and after treatment.
Comparison of clinical parameters of study participants versus associated outcomes for patients on other DC/Imiquimod studies. | Up to 24 Months
  A comparison of whether the clinical parameters associated with outcomes described for patients on other DC/Imiquimod protocols hold for subjects treated on this study.
Estimation of the Proportion of Subjects with Recurrent Pediatric Brian Tumors who are able to complete DC Vaccine therapy and DC Vaccine + Lysate Therapy. | Up to 24 months
  Estimation of the proportion of subjects with recurrent pediatric brain tumors who are able to receive all administrations of DC, and the proportion who are able to receive all administrations of DC and Lysate.
Identification of Parameters Associated with Poorer Activity of the Vaccine in Study Participants | Up to 24 Months
  Identification of parameters associated with poorer activity of the DC Vaccine in Study Participants in order to develop therapies to augment vaccine therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Ziga, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States